CLINICAL TRIAL: NCT04536753
Title: The Utility of Customised Growth Charts for Identifying Macrosomia and the Effect of Intervention
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Other Study IDs: SIMPS01
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-07

CONDITIONS: Obstetric Complication; Ultrasound; Induction of Labor Affected Fetus / Newborn; Fetal Growth Complications
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suspected large for gestational age (LGA): Women with pregnancies suspected to be complicated by fetuses weighing more than the 90th centile on customised growth chart and induced for this reason prior to 287 days as the main indication without diabetes.
  Interventions: Procedure: Induction of labour
- Women with diabetes (DM): Women with diabetes in pregnancy induced at between 259 and 266 days if on treatment and 273 days if gestational diabetes managed with diet alone.
  Interventions: Procedure: Induction of labour
- Control: All other women induced at or after 280 days of gestation
  Interventions: Procedure: Induction of labour

INTERVENTIONS:
Procedure: Induction of labour — Induction of labour using amniotomy, vaginal prostaglandin administration and syntocinon in combination as per protocol.

SUMMARY:
Best management of suspected large for gestational age (LGA) fetuses is unclear. In some hospitals women with an LGA fetus by customised growth charts are are offered earlier induction. This study aimed to examine scan accuracy for this group and the outcome with intervention.

DETAILED DESCRIPTION:
This is a retrospective cohort study of pregnant women taken from 3 groups; women with a suspected LGA fetus (LGA), women with diabetes (DM) and a control group of women that underwent induction of labour at or after 40 weeks. Scan accuracy using GROW and WHO charts in the LGA and DM cohorts was assessed using ROC curves and outcomes between the cohorts was compared.

ELIGIBILITY:
Inclusion Criteria:

* Induced labour of a singleton pregnancy at Northumbria Healthcare Foundation trust resulting in a delivery between 01/01/2018 and 31/12/2018.

Inclusion in the LGA group means that the main indication for induction is recorded as suspected macrosomia.

Inclusion in the Diabetic group means diabetes was pre-existing or arose in pregnancy, diagnosed by oral glucose tolerance testing from 24-30 weeks or by home blood glucose monitoring with standard thresholds as per NICE ng3. Induction had to be undertaken with diabetes as the (co)indication.

Inclusion criteria for the control group was induction of labour at or after 280 days gestation

Exclusion Criteria:

Previous caesarean section Multiple pregnancy Fetal concerns pre-induction: abnormal antenatal trace or abnormal doppler flow studies on antenatal ultrasound

* Cases of induction for suspected LGA are to be excluded if there is a co-indication of obstetric cholestasis, hypertensive disorder or diabetes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women booked for their care at Northumbria Healthcare Trust in North East England: a predominantly white British female population with rates of obesity above the national average.
Sampling Method: Non-Probability Sample
Enrollment: 845 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | through study completion, an average of 1 year
  Caesarean section and assisted delivery rates
Shoulder dystocia rate | through study completion, an average of 1 year
  Any clinically diagnosed cases of shoulder dystocia where the shoulders did not deliver with routine axial traction on the next contraction after the head was delivered.
Estimated blood loss | through study completion, an average of 1 year
  Blood loss as estimated by the clinical team
Obstetric Anal Sphincter Injury | through study completion, an average of 1 year
  Any tear involving the external anal sphincter and/or rectal mucosa
Admission to special care baby unit (SCBU) | through study completion, an average of 1 year
  Admission of neonate to neonatal unit from labour ward
Epidural rate | through study completion, an average of 1 year
  Use of epdiural analgesia intrapartum
Birthweight | through study completion, an average of 1 year
  Neonatal weight as taken following delivery

OTHER OUTCOMES:
Prediction of WHO birthweight >90th centile by scan estimated weight centile on WHO chart | through study completion, an average of 1 year
  As above
Birthweight centile as per customised chart | through study completion, an average of 1 year
  Birthweight centile given birthweight and maternal characteristics as per perinatal institute
Birthweight centile as per WHO population chart | through study completion, an average of 1 year
  Based on Kiserud T, Piaggio G, Carroli G, Widmer M, Carvalho J, et al. (2017) The World Health Organization Fetal Growth Charts: A Multinational Longitudinal Study of Ultrasound Biometric Measurements and Estimated Fetal Weight. PLOS Medicine 14(1): e1002220. https://doi.org/10.1371/journal.pmed.1002220
Scan error as a percentage of estimated fetal weight | through study completion, an average of 1 year
  Difference between birthweight and what it was expected to be based on estimated weight (using perinatal institutes calculator) at scan, given as a percentage of that estimated weight
Prediction of Customised growth chart birthweight >90th centile by estimated weight on scan | through study completion, an average of 1 year
  As above
Prediction of birthweight >4kg based on projected weight at time of delivery from scan estimated weight | through study completion, an average of 1 year
  As above

CONTACTS AND LOCATIONS:
Locations (1):
- Benjamin Simpson, Newcastle upon Tyne, Tyne and Wear, United Kingdom